CLINICAL TRIAL: NCT02899442
Title: Cardiovascular Risk Prevention Among Night Workers
Acronym: Heart-Of-Night
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: assistance of the French National Health Insurance Fund for Employees (CNAMTS) (Unknown); French Directorate General of Health (DGS) (Unknown); ARC Foundation for Cancer Research (Other); National Cancer Institute, France (Other Government); French National Institute for Prevention and Education in Health (INPES) (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); French Inter-Departemental Agency for the Fight against Drugs and Addictive Behaviors (Mildeca) (Unknown); French Social Security Scheme for Liberal Professionals (RSI) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC31/14/7341; 2015-A00895-44 (Other: ID-RCB)
Record Dates: First submitted 2016-09-02; First posted 2016-09-14 (Estimated); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Cardiovascular Diseases
Keywords: cardiovascular risk; Occupational Health; night work; Public Health; Preventive Health Services
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Workplace

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- individual prevention (No Intervention): The individual preventive advice will be delivered to the control group by occupational physicians during routine medical examinations (defined by law, each 6 months), in occupational medical centres. The type and time spent to explain this advice will be collected in case report form.
  To ensure each night workers included in the control group received the same advice, a booklet was provided outlining the content under 5 main headings:
  1. Information about health risks for night workers
  2. Dietetic intake
  3. Leisure physical activities
  4. Sleep and alertness
  5. Lifestyle behaviors (Tobacco, alcohol and psychoactive drugs consumption)
  That's a current practice in France for Occupational physicians.
- individual and collective prevention (Experimental): In addition to this individual prevention, the night workers from the experimental group will benefit from implementation of preventive actions in the workplace (collective prevention in workplace ). These collective preventive measures will be dispensed by the occupational health team (occupational physicians and technician of occupational risks prevention).
  Interventions: Other: collective prevention in workplace

INTERVENTIONS:
Other: collective prevention in workplace — From countermeasures referenced in guidelines, some tools were also created by the committee to standardize all preventive actions and to define measurable indicators. A specific monitoring for checking their applicability and for evaluating the duration of implementation is planned.Collective actions are classified in 7 categories:1)Standardized information of night work risk on health and countermeasure to prevent them, 2)Acknowledgement of the existence of the risk, thereby helping to raise general awareness, 3)Improvement of characteristics of night work (rhythm, rest, time to start and to end, schedule forecasted, duration of night work),4)Improvement of related conditions at night work (Job strain, monotonous or repetitive tasks, manager's help, collective co-operation; Light environment; Occupational physical activities, 5)Sleep improvements ,6)Improvement of dietetic intakes at work, 7)Improvement of leisure physical activity's practice within the work site
  Arms: individual and collective prevention

SUMMARY:
With around 15 to 20% of workforce engaging in nightshift work in modern society for obvious economic and social reasons, the consequences of night work on cardiovascular risks are substantial. Compared to day workers, it was reported higher risks of cardiovascular diseases (estimated at 40%) and of metabolic syndrome (1.5 times) in shift workers. The occurrence of metabolic syndrome increases the risk to develop high blood pressure, diabetes and cardiovascular events. Because some characteristics of night work are potentially modifiable, some preventive strategies could be applied to reduce its adverse effects. For shift workers, some recent guidelines (High Health Authority, 2012 & 2016) and fruitful literature propose to develop regular assessments of cardiovascular risk factors and occupational activities, and stress the need to expand preventive strategies. Moreover, some recent French laws provide an opportunity to implement preventive interventions and specific monitoring through the occupational physicians network. However, whether the concept is defined, the exact content, method and the potential benefits are unknown. The investigator assume that individual advice related to collective countermeasures referenced on guidelines (applied on worksite within plant) could lead a better improvement on incidence of metabolic syndrome compared to those that benefit only individual advice.

Main objective:

To measure the benefit from implementation of individual and collective prevention (dispensed in worksites within plants) on metabolic syndrome compared to strategy relying only on individual prevention among night workers, over 2 years' follow-up. The secondary objectives of the study are to evaluate in both groups:

1. Observance of different types of preventive strategies
2. Impact of observance of preventive advice on metabolic syndrome in shift workers and on each component of metabolic syndrome
3. Determinants which promote the up-take of preventive strategies among night workers
4. The countermeasures which could be applied and effective within company 5) Medico-economic assessment is planned from an ancillary study.

DETAILED DESCRIPTION:
Among the various causes of mortality, deaths attributable to cardiovascular diseases (CVD) are the most widespread worldwide. Despite major progress being made, the risk remains. Occupational factors such as shift work have emerged as potential CV risk factors. With around 15 to 20% of workforce engaging in nightshift work in modern society for obvious economic and social reasons, the consequences of which on occupational and social inequalities are substantial. Compared to day workers, it was reported higher risks of cardiovascular diseases (estimated at 40%) and of metabolic syndrome (1.5 times) in shift workers. The occurrence of metabolic syndrome increases the risk to develop high blood pressure, diabetes and cardiovascular events. Because some characteristics of night work are potentially modifiable, some preventive strategies could be applied to reduce its adverse effects. For shift workers, some recent guidelines (High Health Authority, 2012) and fruitful literature propose to develop regular assessments of cardiovascular risk factors and occupational activities, and stress the need to expand preventive strategies. Moreover, some recent French laws provide an opportunity to implement preventive interventions and specific monitoring through the occupational physicians network. However, whether the concept is defined, the exact content, method and the potential benefits are unknown. The investigator assume that individual advice related to collective countermeasures referenced on guidelines (applied on worksite within plant) could lead a better improvement on incidence of metabolic syndrome compared to those that benefit only individual advice.

* Research objectives Main objective: To measure the benefit from implementation of individual and collective prevention (dispensed in worksites within plants) on metabolic syndrome compared to strategy relying only on individual prevention among night workers, over 2 years' follow-up. The secondary objectives of the study are to evaluate in both groups: 1) Observance of different types of preventive strategies 2) Impact of observance of preventive advice on metabolic syndrome in shift workers and on each component of metabolic syndrome 3) Determinants which promote the up-take of preventive strategies among night workers 4) The countermeasures which could be applied and effective within company 5) Medico-economic assessment is planned from an ancillary study.
* Methodology This study is designed as a multicenter, cluster randomized interventional controlled trial, to reduce the incidence of metabolic syndrome among night workers. Randomization will be performed on 100 occupational physicians (volunteers to participate), to apply one of both interventions. 3056 volunteers' night workers will be recruited from the employees regularly monitored by each physician during the routine medical monitoring. Two parallel groups will be performed: control group and experimental group. A two-year follow-up will be organized including check-points every 6 months. Control group: Every 6 months (T0, 6, 12, 18 months), standardized preventive individual advice focused on cardiovascular risk in night workers will be delivered by occupational physicians. Experimental group: In addition to this individual advice, preventive interventions dispensed on worksite will be carried out. Counter-measures will be applied by occupational health team to improve working conditions. By using a self-questionnaire, a medical questionnaire, a medical examination, biological sample, and specific follow-up of preventive interventions, the assessments will be performed. Study Primary outcome: Reduction of incidence of metabolic syndrome between the two groups (control and experimental) over 2 years' follow up.

Descriptive analysis according to the clusters and also to the both groups will be provided. Multivariate analysis, according to specific design of study (clusters), will be performed by multilevel analysis or marginal analysis. Given the specificity of self-employed people belonging to 'Regime social des independents, a target population will be added. The medical monitoring and individual prevention will be carried out by occupational physicians from occupational disease centres.

• Expected results From implementation of preventive strategies, investigator will expect: 1) The health improvement among night workers by decreased incidence of metabolic syndrome; by improved quality of life; 2) A improvement of social and professional development of night workers by a better tolerance of night work, and job retention; 3) Behavioral improvement by a positive impact of individual and collective behavioral changes on cardiovascular risks; 4) Practical actions by identifying factors which influence the implementation of preventive actions; 5) By this project, investigator would like also to determine some relevant, practical and effective actions which could be generalized at all night workers in preventive health public Policy.

ELIGIBILITY:
INCLUSION CRITERIA:

* For occupational physicians (cluster level)
* Being volunteer
* Physician is responsible of the night workers' monitoring, in plants with at least 10 employees
* Working in multidisciplinary collaborations (occupational physicians and technician on prevention of occupational risks)
* Carrying out professional activities in the 4 referenced regions.
* Performing medical monitoring of night workers every 6 months in accordance with the legislation, as outlined previously.
* For night workers (subject level) night worker must work in a plant with at least 10 employees
* Have a permanent contract and a stable job during the next 2 years
* Be aged 18 years and older participate voluntarily and agree to sign a consent form

EXCLUSION CRITERIA:

1) Main Exclusion criteria:

* For occupational physicians (cluster level)
* Failing to comply with inclusion criteria
* Having planned giving up occupational activities during next 2 years
* For night workers: (subject level)
* Failing to comply with inclusion criteria
* Failing to speak and/ or understand French language
* Being pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3056 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Change of Metabolic Syndrome Factors | inclusion (T0), and 24 months (T24)
  Measure of Metabolic Syndrome Factors, Reduction of incidence of metabolic syndrome between the two groups (control and experimental) over 2 years' follow up. Metabolic syndrome defined as three or more among the following five criteria are present: 1) waist circumference (≥102 cm for male; ≥ 88 cm for female); 2) plasma triglycerides ≥ 1.7 mmol/l or treatment; 3) HDL cholesterol<1.0 mmol/l for male and 1.3 mmol/l for female or treatment, 4) blood pressure ≥ 130/85 mmHg or treatment; 5) fasting glycaemia ≥ 5.5 mmol/l or treatment 35.

SECONDARY OUTCOMES:
Change of preventive interventions | At inclusion (T0), and 24 months (T24)
  the rate of number of countermeasures needed at baseline by calculated number of countermeasures applied at the end of study; the frequency of countermeasures applied.

CONTACTS AND LOCATIONS:
Overall Officials: Yolande ESQUIROL, MDPhD, Principal Investigator — esquirol.y@chu-toulouse.fr
Locations (1):
- Toulouse University Hospital (CHU de Toulouse), Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided